CLINICAL TRIAL: NCT05627635
Title: A Phase I/II Clinical Trial of FOLFOX Bevacizumab Plus Botensilimab and Balstilimab (3B-FOLFOX) in Patients With MSS Metastatic Colorectal Cancer
Brief Title: FOLFOX and Bevacizumab in Combination With Botensilimab and Balstilimab (3B-FOLFOX) for the Treatment of Microsatellite Stable (MSS) Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22251; NCI-2022-09458 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22251 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-11-17; First posted 2022-11-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colon Adenocarcinoma; Metastatic Colorectal Adenocarcinoma; Metastatic Microsatellite Stable Colorectal Carcinoma; Metastatic Rectal Adenocarcinoma; Stage IV Colon Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — balstilimab; Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Fluorouracil; dehydroftorafur; Leucovorin; Magnetic Resonance Spectroscopy; Oxaliplatin; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I (3B-FOLFOX) (Experimental): Patients receive FOLFOX, bevacizumab, balstilimab, and botensilimab IV on study. Patients undergo an x-ray, CT scan, PET scan, and/or MRI throughout the trial. Patients also undergo blood sample collection during screening and on study.
  Interventions: Biological: Balstilimab; Biological: Bevacizumab; Procedure: Biospecimen Collection; Biological: Botensilimab; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Procedure: Positron Emission Tomography; Procedure: X-Ray Imaging
- Phase II, Arm I (3B-FOLFOX) (Experimental): Patients receive FOLFOX, bevacizumab and balstilimab IV with botensilimab IV at a lower dose on study. Patients undergo an x-ray, CT scan, PET scan, and/or MRI throughout the trial. Patients also undergo blood sample collection during screening and on study.
  Interventions: Biological: Balstilimab; Biological: Bevacizumab; Procedure: Biospecimen Collection; Biological: Botensilimab; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Procedure: Positron Emission Tomography; Procedure: X-Ray Imaging
- Phase II, Arm II (3B-FOLFOX) (Experimental): Patients receive FOLFOX, bevacizumab and balstilimab IV with botensilimab IV at a higher dose on study. Patients undergo an x-ray, CT scan, PET scan, and/or MRI throughout the trial. Patients also undergo blood sample collection during screening and on study.
  Interventions: Biological: Balstilimab; Biological: Bevacizumab; Procedure: Biospecimen Collection; Biological: Botensilimab; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Procedure: Positron Emission Tomography; Procedure: X-Ray Imaging

INTERVENTIONS:
Biological: Balstilimab — Given IV
  Other Names: AGEN 2034; AGEN-2034; AGEN2034
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Zirabev
Procedure: Biospecimen Collection — Undergo a blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Botensilimab — Given IV
  Other Names: AGEN 1181; AGEN-1181; AGEN1181; Anti-CTLA-4 Monoclonal Antibody AGEN1181
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Procedure: Positron Emission Tomography — Undergo a PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: X-Ray Imaging — Undergo an x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Radiographic Imaging; Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase I/II trial tests the safety, side effects, best dose, and efficacy of FOLFOX and bevacizumab in combination with botensilimab and balstilimab (3B-FOLFOX) in treating patients with microsatellite stable (MSS) colorectal cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Chemotherapy drugs, such as FOLFOX, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Balstilimab and botensilimab are in a class of medications called monoclonal antibodies. They bind to proteins, called PD-L1 and CTLA-4, which is found on some types of tumor cells. These PD-1 and CTLA-4 proteins are known to affect the body's defense mechanism to identify and fight against tumor cells. The combination of these drugs may lead to improved disease control and outcomes in patients with MSS metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of leucovorin calcium, fluorouracil, oxaliplatin (FOLFOX) bevacizumab, balstilimab and botensilimab at each dose level in order to inform the recommended phase 2 dose (RP2D). (Phase I) II. To assess the overall response rate of FOLFOX bevacizumab, balstilimab at 240 mg and botensilimab at 25 mg and 75 mg (depending on dose level). (Phase II)

SECONDARY OBJECTIVES:

I. To assess the overall response rate, progression-free survival (PFS), and overall survival (OS) of FOLFOX bevacizumab, balstilimab at 240 mg and botensilimab at 25 mg and 75 mg (depending on dose level). (Phase I) II. To estimate the median PFS and median OS associated with FOLFOX bevacizumab, balstilimab at 240 mg and botensilimab at 25 mg and 75 mg botensilimab (depending on dose level). (Phase II) III. To estimate the duration of response associated with FOLFOX bevacizumab, balstilimab at 240 mg and botensilimab at 25 mg botensilimab and 75 mg (depending on dose level). (Phase II) IV. To evaluate the safety/feasibility of FOLFOX bevacizumab, botensilimab, and balstilimab, through the assessment of adverse events. (Phase II) V. To describe the rate of secondary resection in all arms of treatment and summarize their outcome in terms of disease relapse post-surgery. (Phase II)

CORRELATIVE OBJECTIVE:

I. Evaluate potential circulating biomarkers of response, resistance, activity, and toxicity.

OUTLINE: This is a phase I, dose-escalation study of botensilimab followed by a randomized phase II study.

PHASE I: Patients receive FOLFOX, bevacizumab, balstilimab, and botensilimab intravenously (IV) on study. Patients undergo an x-ray, computed tomography (CT) scan, positron emission tomography (PET) scan, and/or magnetic resonance imaging (MRI) throughout the trial. Patients also undergo blood sample collection during screening and on study.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive FOLFOX, bevacizumab and balstilimab IV with botensilimab IV at a lower dose on study. Patients undergo an x-ray, CT scan, PET scan, and/or MRI throughout the trial. Patients also undergo blood sample collection during screening and on study.

ARM II: Patients receive FOLFOX, bevacizumab and balstilimab IV with botensilimab IV at a higher dose on study. Patients undergo an x-ray, CT scan, PET scan, and/or MRI throughout the trial. Patients also undergo blood sample collection during screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 1
* Life expectancy >= 3 months
* Patients should have a pathologically proven diagnosis of colorectal adenocarcinoma
* Histological or cytological confirmed microsatellite stable (MSS) adenocarcinoma of colon or rectum. Microsatellite status should be performed per local standard of practice (immunohistochemistry [IHC] and or polymerase chain reaction [PCR], or next-generation sequencing, the presence of POLE mutations will be collected if available through next-generation sequencing)
* Patients should have measurable metastatic disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines
* Patients should not have a history of perforations or fistulas
* For the safety cohorts (phase I): Metastatic colorectal cancer with 0 to 2 prior lines of therapy prior to enrollment on study and without prior progression within 3 months from last dose of oxaliplatin, in the event of prior oxaliplatin exposure. Evidence of radiographic progression after last treatment before enrollment should be documented

  * Patients with prior FOLFOX therapy should not have required dose modifications and should not have experienced unacceptable toxicities
  * Patients with other prior 5-FU-based therapies should not have required prior fluorouracil (5-FU) dose modifications below 2400 mg/m^2 every 2 weeks
  * No prior oxaliplatin hypersensitivity
  * 4 weeks should have elapsed from last prior chemotherapy and initiation of study treatment
* For the efficacy cohorts (phase II): No prior treatment for metastatic disease. If prior FOLFOX adjuvant therapy was administered, there should be no evidence of disease relapse within the first 12 months after completion of adjuvant therapy
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (within 7 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 2.5 x ULN, unless presence of liver metastases for which =< 5 x ULN is allowed (within 7 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 2.5 x ULN, unless presence of liver metastases for which =< 5 x ULN is allowed (within 7 days prior to day 1 of protocol therapy)
* Creatinine clearance >= 40 ml/min (within 7 days prior to day 1 of protocol therapy)
* Alkaline phosphatase =< 3 x ULN (within 7 days prior to day 1 of protocol therapy)
* Hemoglobin >= 9 g/dl (within 7 days prior to day 1 of protocol therapy)
* Absolute neutrophil count (ANC) >= 1500/ul (within 7 days prior to day 1 of protocol therapy)
* Platelets >= 100,000/mm^3 (within 7 days prior to day 1 of protocol therapy)
* Albumin >= 3.0 g/dl (within 7 days prior to day 1 of protocol therapy)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (within 7 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
  * Females of non-childbearing potential defined as:

    * >= 50 years of age and has not had menses for greater than 1 year
    * Amenorrheic for >= 2 years without a hysterectomy and bilateral oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation
    * Status is post-hysterectomy, bilateral oophorectomy, or tubal ligation
* Women patients of reproductive potential must use effective contraception while receiving oxaliplatin and for 9 months after the final dose. Men with female partners of reproductive potential must use effective contraception while receiving oxaliplatin and for 6 months after the final dose. If patients discontinue oxaliplatin more than 9 months (females) or 6 months (males) before discontinuation of balstilimab and/or botensilimab, females and males of childbearing potential must use an effective method of birth control or abstain from sexual activity for the course of the study through at least 90 days after the last dose of balstilimab and/or botensilimab

Exclusion Criteria:

* Prior immunotherapy
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Prior allogeneic organ transplantation
* Surgical intervention within 4 weeks prior to study treatment, except for minor procedures such as port placement
* Prior allergic reaction or hypersensitivity to any of the study drug components
* Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years before starting treatment, i.e., with use of disease-modifying agents or immunosuppressive drugs
* Uncontrolled hypertension, defined as systolic blood pressure (SBP) >150, diastolic blood pressure (DBP) > 90
* History of acute thrombotic venous events in the last 30 days before enrollment. If within 30 days, the patient should be on anticoagulants and without symptoms
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 12 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class >= III), or serious uncontrolled cardiac arrhythmia requiring medication
* Obstructive bowel symptoms related to unresected primary or carcinomatosis
* Any persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] grade >= 2) from prior cancer therapy, excluding endocrinopathies stable on medication, stable neuropathy that is grade 1 or less, and alopecia
* Non-healing wounds
* Symptomatic active bleeding
* Grade >= 2 proteinuria as demonstrated by >= 2+ protein and >= 1.0 g of protein with 24-hour urine collection (patients found to have >= 2+ protein on dipstick urinalysis must have 24-hour urine collection and demonstrate < 1 g of protein in 24 hours in order to be eligible for the study)
* Active brain metastases or leptomeningeal metastases with the following exceptions:

  * Treated brain metastases require a) surgical resection, or b) stereotactic radiosurgery. These patients must be off steroids >= 10 days prior to randomization for the purpose of managing their brain metastases. Repeat brain imaging following surgical resection or stereotactic radiosurgery at least 4 weeks from treatment should document lack of progression
* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to the first dose of study treatment, i.e., patients with a history of prior malignancy are eligible if treatment was completed at least 2 years before the first dose of study treatment and the patient has no evidence of disease. Patients with history of prior early-stage basal/squamous cell skin cancer, low-risk prostate cancer eligible for active surveillance or noninvasive or in situ cancers who have undergone definitive treatment at any time are also eligible
* Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* History or current evidence of any condition, co-morbidity, therapy, any active infections, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Known previous severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to cycle 1 day 1 (C1D1)
* Uncontrolled infection with human Immunodeficiency virus (HIV). Patients on stable highly active antiretroviral therapy (HAART) with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required
* Known to be positive for hepatitis B virus (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection. Patients who are receiving or who have received anti-HBV therapy and have undetectable HBV deoxyribonucleic acid (DNA) for at least 6 months prior to study entry are eligible. Serological testing for HBV at screening is not required
* Known active hepatitis C virus (HCV) as determined by positive serology and confirmed by polymerase chain reaction (PCR). Patients on or who have received antiretroviral therapy are eligible provided they are virus-free by PCR for at least 6 months prior to study entry. Serological testing for HCV at screening is not required
* Grade 2 or above neuropathy at the time of enrollment
* Dependence on total parenteral nutrition or intravenous hydration
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (phase I) | Up to 6 weeks
  Toxicity, graded according to the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. A dose limiting toxicity is a toxicity that occurs in the first 6 weeks of treatment with 3B-FOLFOX and that is attributed at least as possibly related to the study drugs
Overall response (phase II) | Up to 5 years
  As assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Will examine the proportion of the liver metastasis among the 60 enrolled patients and carry out subgroup analysis for overall response for patients with and without liver metastasis.

SECONDARY OUTCOMES:
Overall response (phase I) | Up to 5 years
  Assessed by RECIST v 1.1. Will examine the proportion of the liver metastasis among the 60 enrolled patients and carry out subgroup analysis for overall response for patients with and without liver metastasis.
Progression-free survival (PFS) (phase I) | Time to disease progression/ relapse or death as a result of any cause, assessed up to 5 years
  Kaplan-Meier curve will be used to assess the PFS. Median survival and the 95% confidence interval (CI) will be reported. The effect of the higher botensilimab dose (75mg versus [vs] 25mg) will be estimated by the hazard ratio (HR) in a Cox proportional hazard model with and without adjustment for clinically relevant covariates. Will examine the proportion of the liver metastasis among the 60 enrolled patients and carry out subgroup analysis for PFS for patients with and without liver metastasis.
Overall survival (OS) (phase I) | Time to death as a result of any cause, assessed up to 5 years
  Kaplan-Meier curve will be used to assess the OS. Median survival and the 95% CI will be reported. The effect of the higher botensilimab dose (75mg vs 25mg) will be estimated by the HR in a Cox proportional hazard model with and without adjustment for clinically relevant covariates. We will examine the proportion of the liver metastasis among the 60 enrolled patients and carry out subgroup analysis for OS for patients with and without liver metastasis.
PFS (phase II) | Time to disease progression or death as a result of any cause, assessed up to 5 years
  Kaplan-Meier curve will be used to assess the PFS. Median survival and the 95% CI will be reported. The effect of the higher botensilimab dose (75mg vs 25mg) will be estimated by the HR in a Cox proportional hazard model with and without adjustment for clinically relevant covariates. Will examine the proportion of the liver metastasis among the 60 enrolled patients and carry out subgroup analysis for PFS for patients with and without liver metastasis.
OS (phase II) | Time to death as a result of any cause, assessed up to 5 years
  Kaplan-Meier curve will be used to assess the OS. Median survival and the 95% CI will be reported. The effect of the higher botensilimab dose (75mg vs 25mg) will be estimated by the HR in a Cox proportional hazard model with and without adjustment for clinically relevant covariates. We will examine the proportion of the liver metastasis among the 60 enrolled patients and carry out subgroup analysis for OS for patients with and without liver metastasis.
Duration of response (phase II) | Time to progression or death, starting at the time when a response is experienced, assessed up to 5 years
Incidence of adverse events (phase II) | Up to 5 years
  Toxicity, graded according to the NCI-CTCAE v5.0.
Surgical resection (phase II) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marwan G Fakih, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States